CLINICAL TRIAL: NCT03650647
Title: Randomized Clinical Trial Comparison of Conventional Versus Conservative Caries Removal in Primary Teeth: a Two-year Evaluation
Brief Title: Comparison of Conventional Versus Conservative Caries Removal in Primary Teeth
Acronym: Caries_removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Apoena de Aguiar Ribeiro, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ARibeiro
Record Dates: First submitted 2018-08-21; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Dental Caries Extending Into Dentin
Keywords: Dental caries; Dentin; Pulp exposure prevention; Deep caries lesion; Conservative Treatment
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Tooth receive one of the two test treatments: Stepwise Excavation (conservative treatment 1), Selective caries removal (conservative treatment 2) and are evaluated in parallel against a control group (indirect pulp capping treatment).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Indirect Pulp Capping (Active Comparator): Nonselective removal to hard dentine (formerly complete excavation or complete caries removal) : removal of soft dentin, only hard dentine is left on the cavity, so that demineralized dentine "free" of bacteria is completely removed.
  Intervention: Total soft and leathery caries removal. Carious dentin removal
  Interventions: Procedure: Carious dentin removal
- Stepwise excavation (Experimental): Stepwise removal is carious tissue removal in 2 stages, i.e., visits. Soft carious tissue is left over the pulp in the first step, while peripheral dentine is prepared to hard dentine to allow a complete and durable seal of the lesion. A provisional restoration is placed, which should be sufficiently durable to last up to 6 months to allow changes in the dentine and pulp to take place. After this period, a second excavation is done and, if there is hard dentin formed, the tooth is restored.
  Intervention: Part of the soft caries is removed. Final restoration is placed on the second visit. Carious dentin removal
  Interventions: Procedure: Carious dentin removal
- Selective caries removal (Experimental): Selective caries removal: only part the soft dentine is removed, so soft carious tissue is left over the pulp, while peripheral enamel and dentine are prepared to hard dentine, to allow a tight seal and placement of a durable restoration.
  Intervention: Part of the soft caries is removed. Final restoration is place over the soft dentin. Carious dentin removal
  Interventions: Procedure: Carious dentin removal

INTERVENTIONS:
Procedure: Carious dentin removal — Carious tissue removal and managing deep cavitated carious lesions in primary teeth.
  Other Names: Indirect Pulp Capping; Stepwise excavation; Selective caries removal

SUMMARY:
The sample will be, at least, 90 primary molars, randomly distributed into three groups: Group 1: IPC; Group 2: SE; Group 3: SCR. Teeth must present deep caries lesions (at least 2/3 of dentin depth), pulp vitality (no clinical or radiographical signs of pulp disease, such as abcesses, fistulae, root resorption, abnormal tooth mobility). This study received approval by the Ethics Committee of Fluminense Federal University (UFF; Brazil) - # CAAE: 58812816.8.0000.5626. The study started in January, 2017; and will finish in December, 2020. Patients will be selected from the public schools in Nova Friburgo. The dental exams and treatment procedures will be done at the clinics from the

School of Dentistry, Health Institute of Nova Friburgo (ISNF). Laboratory proceedings will be done at:

* Clinical and Microbiological Research Laboratory (LAB PECMA - ISNF) - Sample storage, bacterial cultivation and identification.
* University of North Carolina at Chapel Hill
* Rio de Janeiro Federal University

DETAILED DESCRIPTION:
The aims of this Randomized Clinical Trial are:

1. to evaluate the risk of pulpal exposure and tooth vitality maintenance of primary molars with deep caries lesions, treated with conservative techniques, such as Stepwise Excavation (SE) or Selective Caries Removal (SCR), and to compare with those teeth treated with Indirect Pulp Capping (IPC);
2. to verify changes in the cultivable microbiota isolated in the deep carious dentin lesions of deciduous molars, before and after performing the procedures of SE;
3. to clinically evaluate dentin reactions to the SE;
4. to provide longitudinal monitoring of changes in the non-cultivable microbiota (microbiome), found in dentin carious lesions of deciduous and permanent molars, compared to the treatments performed;
5. to determine, in vitro, the microbial metabolome of different strains isolated from dentin samples under conditions of high and low cariogenic challenge;
6. to correlate, in vitro, the microbial metabolites with the clinical classification of the cavitated lesions from which these samples originated.

The sample will be, at least, 90 primary molars, randomly distributed into three groups: Group 1: IPC; Group 2: SE; Group 3: SCR. Teeth must present deep caries lesions (at least 2/3 of dentin depth), pulp vitality (no clinical or radiographical signs of pulp disease, such as abcesses, fistulae, root resorption, abnormal tooth mobility). This study received approval by the Ethics Committee of UFF (Brazil) - # CAAE: 58812816.8.0000.5626. The study started in January, 2017; and will finish in December, 2020. Patients will be selected from the public schools in Nova Friburgo. The dental exams and treatment procedures will be done at the clinics from the

School of Dentistry, Health Institute of Nova Friburgo (ISNF). Laboratory proceedings will be done at:

LAB PECMA - ISNF - Sample storage, bacterial cultivation and identification University of North Carolina at Chapel Hill Rio de Janeiro Federal University

ELIGIBILITY:
Inclusion Criteria:

1. The child need to be healthy;
2. This should be in the age range of 4 to 6 years of age;
3. The primary molars to be submitted to treatment should have the following characteristics: deep caries lesion (greater than or equal to 2/3 of dentine thickness) without clinical or radiographic aspects of pulp lesion, restoration margins above gingival line, absence of spontaneous pain or mobility, absence of periodontal changes, roots compatible with pulpal maturation stage.

Exclusion Criteria:

1. Children under use of controlled drugs or antibiotics.
2. Children who presented with some neurological or motor disorder that could influence the treatment procedure.
3. Molars with more than three lost walls or margins in subgingival area.
4. Patients with allergies to the medications used.
5. Patients in the pulpal regression stage in which the tooth is likely to be lost within 12 months.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2020-01-05 (Estimated)

PRIMARY OUTCOMES:
Pulp vitality maintenance diagnosed by clinical exam | Through study completion, up to three years.
  Among the three treatment protocols, which one will have better prognosis in maintaining pulp vitality. The clinical parameters of pulpal failures are: pain, presence of abscess, fistulae and/or abnormal tooth mobility.
Pulp vitality maintenance diagnosed by radiograph exam | Through study completion, up to three years.
  The prognosis of maintaining pulp vitality will be acessed by radiological signs of loss of vitality, as presence of abnormal root resorption and/or bone resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Apoena A Ribeiro, PhD, Principal Investigator — University of North Carolina, Chapel Hill